CLINICAL TRIAL: NCT02818270
Title: Evaluation of Aerosolized Drugs Deposition Delivered Through a Mechanical Ventilator
Brief Title: Evaluation of Aerosolized Drugs Deposition During Mechanical Ventilation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung University (Other)
Collaborators: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Hui-Ling Lin, Assistant professor, Chang Gung University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: NMRPD1E0911
Record Dates: First submitted 2016-06-20; First posted 2016-06-29 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2017-01

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Albuterol; Acetylcysteine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Drug depositions (Experimental): Aerosol drug deposited delivered on the inhaled and exhaled filters and protective filters were evaluated. Salbutamol and Acetylcysteine were delivered by a jet nebulizer through a mechanical ventilator.
  Interventions: Drug: Salbutamol; Drug: Acetylcysteine

INTERVENTIONS:
Drug: Salbutamol — Salbutamol (albuterol ) was delivered by a jet nebulizer with a 50 pis oxygen flow at 6 L/min.
  Other Names: albuterol
Drug: Acetylcysteine — Acetylcystine was delivered by a jet nebulizer with a 50 pis oxygen flow at 6 L/min.
  Other Names: Mucomyst

SUMMARY:
Aerosol delivery through a ventilator is influenced by numerous factors from ventilator-related, circuit-related to device-related factors. Aerosolized drug delivery through a ventilator system was studied on bench model with albuterol, yet the results were often overestimated. The objective of this study was to evaluate inhaled bronchodilator and mucolytic agents delivered through a ventilator system.

DETAILED DESCRIPTION:
Aerosolized medication is used widely to patients with respiratory illness and admitted in the intensive care unit, and includes bronchodilators, steroids, mucolytics, and antibiotics. Aerosol delivery through a ventilator is influenced by numerous factors from ventilator-related, circuit-related to device-related factors. Aerosolized drug delivery through a ventilator system was studied on bench model with albuterol, yet the results were often overestimated. Only few clinical trials on aerosol delivery deposition were published in the last decades. In addition, inhaled bronchodilators, mucolytics, antibiotics, and steroids are often administered to ventilated patients in the intensive care units in Taiwan, but they are never studied. Therefore, the aim of this study was to evaluate inhaled bronchodilator and mucolytics (acetylcystine) delivered by a jet nebulizer through a ventilator system to intubated patients.

ELIGIBILITY:
Inclusion Criteria:

* Mechanical ventilated patients with an endotracheal tube intubated
* Receiving aerosol therapy with salbutamol or acetylcystine
* On relatively stable medical condition

Exclusion Criteria:

* Pregnant
* Unstable hemodynamic status (e.g. blood pressure <100/60 mmHg, under Intra-aortic balloon pump)
* Infected with airborne pathogens (e.g. tuberculosis or Influenza virus)
* Poor oxygenation (fraction of inspiratory oxygen >0.8, under high frequency oscillatory ventilation, or extracorporeal membrane oxygenation)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Inhaled drug dose | Inhaled drug dose was collected Immediately after each nebulization, expected average of 20 minutes
  Drug depositions in inspiratory filters were analyzed by a spectrophotometer.

SECONDARY OUTCOMES:
exhaled drug dose | Exhaled drug dose was collected Immediately after each nebulization, expected average of 20 minutes
  Drug depositions in expiatory filters were analyzed by a spectrophotometer.

CONTACTS AND LOCATIONS:
Overall Officials: Hui-Ling Lin, MSc, Principal Investigator — Chang Gung University
Locations (1):
- Chiayi Chang Gung Memorial Hospital, Chiayi City, Taiwan

IPD SHARING:
Plan to Share IPD: No